CLINICAL TRIAL: NCT00558961
Title: A Phase I-II Trial of Gleevec (Imatinib Mesylate) in Combination With Chlorambucil in Previously Treated Chronic Lymphocytic Leukemia (CLL) Patients
Brief Title: Dose Escalation Study of Gleevec and Chlorambucil in Previously Treated Chronic Lymphocytic Leukemia Patients
Acronym: GL-CLB-001
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unsatisfactory enrollment
Sponsor: Jewish General Hospital (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Sarit Assouline, Associate Professor, Department of Oncology, McGill University, Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR0506PI; REC:05-054
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; chronic lymphocytic leukemia; leukemia; gleevec; chlorambucil
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — Imatinib Mesylate; Chlorambucil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental): Gleevec Chlorambucil
  Interventions: Drug: Gleevec and Chlorambucil

INTERVENTIONS:
Drug: Gleevec and Chlorambucil — The first cohort will receive Gleevec at 300 mg daily on days 1-10 and chlorambucil 8mg/m2/d from day 3-7. This will be repeated every 28 days. Cohort 2 will receive 400 mg Gleevec and Cohort 3 will receive 600 mg Gleevec. Each dose level may be expanded up to 6 patients if 1 of 3 patients experiences any dose limiting toxicities.
  Other Names: Gleevec (imatinib mesylate); Chlorambucil

SUMMARY:
The purpose of this study is to determine maximum tolerated dose of Gleevec in combination with Chlorambucil in previously treated CLL patients.

DETAILED DESCRIPTION:
A recent study by Aloyz et al demonstrated a synergistic effect of imatinib on chlorambucil-mediated cytotoxicity in CLL cells in vitro. Imatinib inhibits c-abl and sensitizes cells to chlorambucil. The Phase I component of the study will determine the maximum tolerated dose and recommended Phase II dose of Gleevec when used in combination with chlorambucil. Once the maximum tolerated dose has been determined, a total of 16 patients will be enrolled in the Phase II component of the study. This study will determine the dose limiting toxicities, pharmacokinetics and pharmacodynamics of Gleevec in combination with chlorambucil.

ELIGIBILITY:
Inclusion Criteria:

* B-cell chronic lymphocytic leukemia (a) Rai stage 0-II with indication for treatment by NCI Working Group Criteria: or (b) Rai stage III or IV.
* Received a minimum of one prior chemotherapy regimen. Prior treatment with corticosteroids, immunotherapies, monoclonal antibodies or radiation therapy is permitted.
* White blood cell count > 25 x 10^9/L
* ECOG 0, 1,or 2.
* Adequate renal and hepatic function
* Platelets > 75 x 10^9/L, transfusion independent.
* Neutrophils > 1.0 x 10^9/L, transfusion independent

Exclusion Criteria:

* Documented prolymphocytic leukemia (PLL; prolymphocytes, 55% in blood)
* Active cardiovascular disease as defined by NYHA class III-IV categorization.
* Intercurrent illness or medical condition precluding safe administration of ribavirin.
* Concurrent use of chronic steroids, except as replacement therapy for adrenal insufficiency
* Known infection with HIV, Hepatitis B or C.
* Concurrent malignancy (other than resected basal or squamous cell skin cancers or in-situ carcinoma).
* Received any previous therapy for CLL within 28 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Measure number of patients at maximum tolerated dose of Gleevec in combination with chlorambucil | 1 month

SECONDARY OUTCOMES:
Report adverse events as a measure of safety | 6 months
Report response to treatment as a measure of efficacy | 6 months
Report level of gleevec concentration at different doses as a measure of pharmacokinetics | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Sarit Assouline, MD, Principal Investigator — Jewish General Hospital; Lawrence Panasci, MD, Study Director — Jewish General Hospital
Locations (2):
- Canada (2):
  - Charles Lemoyne Hospital, Greenfield Park, Quebec
  - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Background] Aloyz R, Grzywacz K, Xu ZY, Loignon M, Alaoui-Jamali MA, Panasci L. Imatinib sensitizes CLL lymphocytes to chlorambucil. Leukemia. 2004 Mar;18(3):409-14. doi: 10.1038/sj.leu.2403247. PMID 14712290